CLINICAL TRIAL: NCT03352401
Title: Gastric Assessment in Ambulatory Surgery : a Prospective Study
Brief Title: Gastric Assessment Ambulatory Surgery
Acronym: GAAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0289
Record Dates: First submitted 2017-11-16; First posted 2017-11-24 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Full Stomach
Keywords: Pulmonary aspiration, full stomach, gastric content inhalation, Mendelson syndrom

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasouund assessment of gastric contents — A qualitative and quantitative ultrasound evaluationof the stomach will be performed when the patient arrives in the pre-anesthesia room. The examination will be held in the right lateral decubitus with a low frequency convex ultrasound probe.

SUMMARY:
The surgical procedures in outpatient surgery are in perpetual increase. However, the peri operative stress can reduce the gastric emptying. A patient's compliance for following the fasting rules cannot be controlled at home. Ambulatory surgery is currently proposed to fragile patients with many comorbidities known to slow gastric emptying. In day case surgery the airway management are often managed with supraglottic device ( laryngeal mask). This device does not protect the respiratory tract and may expose the patient to a risk of inhalation of gastric content (if not empty).

This study aim to mesure the prevalence of full stomachs in outpatient surgery and to observe any changes in anesthetic management secondary to the ultrasound assessment of gastric content. It will confront theoretical full stomach risk factors with ultrasound findings. The practical and clinical relevance of such a technique in the context of outpatient surgery will be assessed in this study. The ultimate goal is to improve the safety of the patient's anesthetic management by controlling the risk of pulmonary aspiration.

DETAILED DESCRIPTION:
Patients will be included during the pre-anesthetic evaluation. The theoretical full stomach risk factors and the anesthetic management will be recorded in the computerized pre-anesthetic evaluation.

A qualitative and quantitative ultrasound evaluation will be performed when the patient arrives in the pre-anesthesia room. The examination will be performed in the right lateral decubitus with a low frequency convex ultrasound probe.

The main objective is to measure the prevalence of patients with a "full stomach" based on ultrasound criteria.

The primary endpoint is the presence of solid or fluid greater than 1.5 ml / kg of the predicted ideal body weight during ultrasonographic evaluation of gastric contents. In this situation, the patient will be considered at high risk of inhalation (considered full stomach).

This study will observe and record any anesthetic changes (ie : airway management) secondary to this ultrasouund assessment of gastric contents.

ELIGIBILITY:
Inclusion Criteria:

Affiliation to social security. Be over 18 years old. Have signed informed consent for this study. Score from the American Society of Anesthesiology (ASA) 1, 2, or 3. Being admitted for ambulatory day care surgery.

Exclusion criteria:

Patients who are protected or unable to give consent Patients with cognitive dysfunction, or unable to give their consent according Pregnant or lactating women. Vulnerable people. Patients with a history of esophageal or gastric surgery Patients suffering from hiatal hernia with esophageal reflux

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ultrasouund assessment of gastric contents : prevalence of patients with a "full stomach" based on ultrasound criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
The prevalence of patients with a "full stomach" based on ultrasound criteria. | one hour
  The presence of solid or fluid greater than 1.5 ml / kg of the predicted ideal body weight during ultrasonographic evaluation of gastric contents.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BIBOULET, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC